CLINICAL TRIAL: NCT06217809
Title: EmpowHer is Prevention Curriculum for Youth Ages 10-15 Years.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alternatives For Girls (Other)
Responsible Party: Principal Investigator, Celia Thomas, Principal Investigator, Alternatives For Girls
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EmpowHer
Record Dates: First submitted 2023-12-28; First posted 2024-01-23 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Abstinence, Sex
MeSH Terms: conditions — Sexual Abstinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EmpowHer (Experimental): The intervention curriculum is designed to address abstinence, and adulthood preparation topics.
  Interventions: Behavioral: The intervention curriculum addresses sexual activity, abstinence, and adulthood preparation topics.

INTERVENTIONS:
Behavioral: The intervention curriculum addresses sexual activity, abstinence, and adulthood preparation topics. — The intervention is youth-co-led, and targets youth in Detroit, Out-Wayne County or geographically similar areas through a 16-unit curriculum totaling 20 hours. Each participant and their parent/guardian will also receive one individual session with a case planner. Parents will receive 3 hours of parental support group. EmpowHer contains lessons and activities focusing on topics relating to abstinence, and teen pregnancy prevention, focusing on adulthood preparation subjects (APS), such as parent-child communication, adolescent development, healthy life skills, and healthy relationships.

SUMMARY:
Alternatives For Girls (AFG's) EmpowHer curriculum is a program for youth who are 10-15 years of age. The curriculum is youth-co-led, and innovative (using online platforms and digitized presentation of material. EmpowHer addresses four adulthood preparation subjects (APS), such as parent-child communication, healthy relationships, adolescent development, and healthy life skills, and can be implemented as an after-school, in/out-of-school-time program.

ELIGIBILITY:
Inclusion Criteria:

Youth who are 10 -15 years of age at the start of the study and residing in Detroit, Outer-Wayne County or geographically similar areas at the time of enrollment will be eligible to participate in the study.

Exclusion Criteria:

Participants who are currently utilizing other services from Alternatives For Girls (AFG), children of AFG staff and youth participating in other sexual health education programs will not be eligible to participate and will be wait-listed until they are no longer receiving other services from AFG (i.e., after-school programs, summer day camps, mentoring, youth leadership programs, and shelter services). These services are unrelated to the study/sexual health education and do not include EmpowHer or Sassy Science. If siblings were to be enrolled, one would be randomly assigned, and the rest would be allowed to participate in the same group as the study sibling but not counted in the evaluation. This is to prevent possible contamination between conditions.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 552 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Recent sexual activity | At 9-month follow up.
  Do participants in the curriculum model (EmpowHer) show reduced rates of sexual activity at 9-month follow up compared to those in a control curriculum (Sassy Science)?
Abstinence | At 9-month follow up.
  Do participants in the curriculum model (EmpowHer) show increased rates of abstinence at (a) 6-month follow-up, and (b) 9-month follow up compared to those in control curriculum (Sassy Science)?

SECONDARY OUTCOMES:
Healthy relationship knowledge | After 20-hour intervention (at post-test).
  Do participants in the curriculum model (EmpowHer) show increased healthy relationship knowledge at post-test compared to those in a control curriculum (Sassy Science)?

CONTACTS AND LOCATIONS:
Locations (1):
- Alternatives For Girls, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Not sharing.